CLINICAL TRIAL: NCT03237533
Title: Comparative Efficacy of Dexamethasone, Doxycycline, Nystatin and Promethazine With Triamcinolone in Orabase as Symptomatic Treatment of Oral Lichen Planus, A Randomized Controlled Trial
Brief Title: Treatment Modalities of Oral Lichen Planus
Acronym: OLP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Durr-e-Sadaf, Demonstrator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123456789
Record Dates: First submitted 2017-07-29; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Dexamethasone; Doxycycline; Nystatin; Promethazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): in this group patients will be treated with Dexamethasone local application
  Interventions: Drug: Dexamethasone
- Control Group (Active Comparator): in this group patients will be treated with dexamethasone, doxycycline and nystattin
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be applied locally on the lesion
  Other Names: Doxycycline, Nystatin, Promethazine, Triamcinolone Orabase

SUMMARY:
Background: Oral lichen planus (OLP) is a chronic inflammatory mucocutaneous autoimmune disease mainly affecting stratum basal of the epithelium. It is very painful and hamper the daily routine of patients e.g. (talking, drinking, eating, maintaining normal relationships). Different topical treatments have been tried for the symptomatic relief of OLP which include topical corticosteroids (TCSs), topical calcineurin inhibitors (TCIs) retinoids, photochemotherapy; amitryptaline; thalidomide; amlexanox and traditional medicines such as curcumin, selenium-ACE combined with itraconazole, glycyrrhiza glabra and aloe vera. But the exact treatment is still unknown.

Objective: To compare the efficacy of Dexamethasone, Doxycycline, Nystatin and Promethazine cocktail with Triamcinolone as topical treatment of OLP Subjects and Methods: 40 patients of symptomatic OLP will be randomly divided in to study and control group. Study group will be given a cocktail containing dexamethasone, doxycycline, nystatin and promethazine and will be advised to rinse with 1 and half teaspoon of this cocktail 3 times a day for 2 minutes for the period of 8 weeks. Study group is also advised to apply an orabase containing 0.1% triamcinolone on lesions 3 times a day for the period of 8 weeks. The control group will be advised to apply only triamcinolone orabase 3 times a day for 8 weeks.

DETAILED DESCRIPTION:
Introduction Oral lichen planus (OLP) is a chronic inflammatory mucocutaneous autoimmune disease mainly affecting stratum basal of the epithelium. It is T-cell mediated immunological disease that mostly occurs bilaterally on buccal mucosa while tongue and gingiva are other commonly involved sites while palatal mucosa and floor of the mouth are rarely affected (Roopashree MR, 2010, Torrente-Castells et al., 2010, Alves et al, 2010). The prevalence of OLP in general population is 0.1-4% (Sugerman et al., 2002) mainly affecting the middle-aged and elderly people (Ingafou et al., 2006) and female: male ratio 2:1 (Shen et al., 2012).

It has six clinical forms: keratotic, reticular, papular, plaquelike white patches, erosive, atrophic, and bullous (Shen et al., 2012). Reticular and erosive form are most common (Alves et al, 2010). Keratotic reticular, papular, plaque like white patches often present with no complaints (Oczko et al, 2011), while erosive, atrophic, and ulcerative lesions are a painful or present with a burning sensation, and thus make eating, speaking, and swallowing difficult (Thongprasom et al., 2007). Histologically, a subepithelial infiltration in the form of dense band of lymphocytes, increased numbers of intraepithelial lymphocytes and the liquefaction degeneration of basal keratinocytes is seen in OLP (Payeras et al., 2013).

Several predisposing factors have been identified which may cause or progress OLP which include immunity, infection, genetics, stress and endocrine. Recent researches showed an increased activity of prolidase and oxidative stress in OLP patients, causing disturbance in the antioxidant defense system (Batu et al, 2016, Ergun et al, 2011). Although the exact cause is still not clear, facts show that an immunological process is involved in OLP which is activated by an unknown antigen that change the basal keratinocytes of the oral mucosa and these alterations cause the cell immune response to attack the keratinocytes. (Ismail et al., 2007, Payeras et al., 2013). This antigen may be intrinsic or extrinsic, or both. Evidence shows that bacteria can be one of the etiologic factors of OLP. An association has already been found between OLP and infection, such as Ebstein Barr virus, Hepatitis C virus, Helicobacter pylori and Candida Albicans. A study also pointed out the allergy to various antigens coming in direct contact with oral cavity to contribute to the etiology of OLP. (D. Wray, 2000) As the etiology is not known therefore there is no definitive treatment for OLP and the mainstay of therapy for improving the life of these patients is symptomatic topical treatment. Topical treatments which have been tried for the symptomatic OLP include topical corticosteroids (TCSs), including betamethasone, clobetasol, dexamethasone and triamcinolone; topical calcineurin inhibitors (TCIs) such as pimecrolimus, tacrolimus or ciclosporin; retinoids such as tretinoin; photochemotherapy; amitryptaline; thalidomide; amlexanox and traditional medicines such as curcumin, selenium-ACE combined with itraconazole, glycyrrhiza glabra and aloe vera.

In a study both tacrolimus 0.1% ointment and pimecrolimus 1% cream were found equally effective for the treatment of OLP (Vohra et al., 2016). Similarly another study showed that Clobetasol propionate (0.05%) was found more effective than triamcinolone acetonate (0.1%) and tacrolimus orabase (0.03%) for the management of OLP. This study also found that triamcinolone 0.1% is superior to tacrolimus 0.03% in terms of effectiveness for the treatment of OLP.(Sivaraman et al., 2016) According to another study both triamcinolone and curcumin paste were found almost equally effective in reducing the pain and improving the appearance of OLP lesions (Kia et al., 2015). In another study it was concluded that combination of Selenium-ACE, corticosteroid and antifungal is a better treatment regimen for the treatment of erosive ulcerative OLP than a capsule of 100 mg Itraconazole plus dexamethsone mouthwash or dexamethasone alone (Belal, 2015). In another similar study cocktail of clobetasol, ketoconazole and amitryptiline was found more efficacious than diluted dexamethasone, nystatin and Diphenhydramine elixir (Javadzadeh et al, 2008). In a comparative study tacrolimus 0.1% cream was found more effective than 0.05% clobetasol propionate cream in reducing pain and healing of OLP lesions (Hettiarachchi et al., 2016). Both thalidomide and dexamethasone were found almost equally effective in another trail (Wu et al., 2010). In a trail of comperison between amlexanox paste and dexamethasone paste both were found equally effective at the end of 7 days in terms of reduction in clinical signs (erosion) and symptoms like pain and burning sensation (Fu et al., 2012). Some herbal medicines have also been tried like Glycyrrhiza glabra and Aloe vera, in a trail to compare the efficacy of 1% Glycyrrhiza glabra In orabase with 0.1% Triamcinolone Acetonide both were found almost equally effective in reducing the pain and improving the appearance of OLP lesions (Najafi et al., 2016) and in another trail both Aloe Vera Mouthwash and Triamcinolone Acetonide were found almost equally effective in reducing the pain and in reducing the size of OLP lesions (Mansourian et al., 2011) So steroids remained the mainstay of treatment for OLP but evidence points towards the involvement of bacterial and fungal infections in the pathogenesis of OLP as according to a recent study disbiosis was found in the buccal surface mucosa of patients of OLP, as certain bacterial species were found in greater no in buccal mucosa of OLP patients so they concluded that an association exists between bacterial disbiosis of buccal mucosa and OLP (He et al., 2017). Similar studies showed that antibiotics relieved symptoms of OLP effectively (Backman & Jontell, 2007; Carbone et al, 1999). OLP is a disease which reduces the individual's resistance and changes the candida albican's role from commensalism to parasitism which is among the normal flora of oral cavity or candida may secondarily infect the OLP lesions and exacerbate the signs and symptoms (santosh gowdru shivanandappa, 2012). In a study 62% of OLP patients were found allergic to different allergens which come in contact with mucosa in daily life so they found that association exists between OLP and allergy (D. Wray, 2000). According to another study mast cell hyperplasia was seen in OLP patients which suggests their role in pathogenesis of OLP (Ankle R et al, 2007) The most used therapy is TCSs however its effectiveness is limited due to opportunistic oral infections in patients with OLP. Adjunct antibiotic therapies have been used to aid in symptomatic relief and improved response has been observed as compared to TCSs alone. however none of the combined therapies have used antifungal as an additive in their local applications, as candida is one of the opportunistic organisms that colonizes affected sites. Role of allergy mechanisms have also been discussed.

Rationale Evidence of involvement of bacterial and fungal infections and allergy in the pathogenesis of OLP suggests the need for the use of antibiotic, anti fungal and antihistamine for the topical treatment of OLP and there is a gap in literature. That's why current trail is being done to evaluate the efficacy of topical doxycycline, nyastatin and promethazine along with dexamethasone for the symptomatic relief of OLP.

Hypothesis Dexamethasone, Doxycycline, Nystatin and Promethazine combination topical rinse are more effective for the treatment of OLP than Triamcinolone alone Objective To compare the efficacy of Dexamethasone, Doxycycline, Nystatin and Promethazine combination topical rinse with Triamcinolone rinse as topical treatment of Oral Lichen Planus.

Operational Definitions • Oral Lichen Planus: Oral lichen planus (OLP) is a chronic inflammatory mucocutaneous autoimmune disease mainly affecting stratum basal of the epithelium.

Subjects and Methods Study Type Randomized control trail (Parallel arm study). Study Setting Department of Oral Medicine & Diagnosis and Department of Dermatology. Madina Teaching Hospital Faisalabad.

Duration The study will be completed in 3 months after the approval of synopsis. Study Population Patients of oral lichen planus visiting Department of Oral Medicine & Diagnosis and Department of Dermatology. Madina Teaching Hospital Faisalabad.

Sampling Technique Purposive Sampling, (Inclusion/exclusion criteria based)

Sample Selection Inclusion Criteria

1. Histopathologically proven patients of OLP of all age groups complaining of symptoms such as pain, burning sensitivity to hot and spicy food.
2. Who have signed informed consent. Exclusion Criteria

<!-- -->

1. Patients who have taken any medication for OLP within 4 weeks before the start of study.
2. Pregnant and lactating women.
3. History of lichenoid reactions to beta blockers, dapsone, oral hypoglycemics, NSAIDS, pencillamine, phenothiazines, sulfonylureas, gold salts or amalgam fillings.

   Sample Size All consecutive OLP patients will be evaluated according to inclusion/exclusion criteria and at least 32 subjects will be enrolled they will be randomly divided into study and control groups.

   The sample size is calculated by the following formula keeping the power of study equal to 90% and level of significance equal to 0.05. The sample size should be 16 in each group.

   [p1(1 - p1) + p2 (1 - p2)] n = × cp,power (p1 - p2)2 (Whitley and Ball, 2002) Desired Level of Significance = 0.05 P1= proportion 1= 70% (0.7) P2= proportion 2= 30% (0.3) Cp, power = 90% =10.5 Sample size in each group = 16 Randomization Randomization will be done by allowing each patient to pick a sealed envelope from a box containing 40 envelopes of which 20 are of study and 20 are of control group.

   Study Variables Socio-demographic/Medical parameters • Age (years), • Gender (male / female), • Education (no-education / secondary / University), • Income (<10000.00- / 10-20000.00 / >20000.00),

   • Smoking (never / former / current),

   • Systemic conditions (CVD / DM / Hepatic / Rheumatoid Arthritis etc),

   • Medications

   • Oral hygiene habits (brushing, floss, dental visit)

   Oral parameters
   * Dimensions of lesion will be measured by with the help of a UNC-12 probe (HDL® Pakistan).
   * Color of lesion will be recorded by standardized pre and post treatment photographic record.
   * Pain or burning sensation will be evaluated by visual analogue scale (VAS).
   * Clinical response (improvement of lesions and symptoms) will be assessed by criteria given by (Escudier et al., 2007).

   Data Collection Method and Instruments After approval from the ethical review committee, patients will be included in the study. Written informed consent will be obtained from all patients prior to the study as a part of ethical practice. 40 patients of symptomatic OLP will be enrolled in the study after evaluation through punch biopsy and other inclusion and exclusion criteria to compensate the loss to follow up as the actual size calculated from the formula was 32. They will be randomly divided in to study and control group each containing 20 patients. At baseline visit after recording the socio-demographic and oral parameters data the local irritant factors in the oral cavity which can aggravate the OLP will be removed by doing basic oral procedures like scaling and root planning restorations, rounding of sharp cusps and replacement of any ill fitting appliances in both the groups.

   Study group will be given a cocktail containing dexamethasone, doxycycline, nystatin and promethazine and will be advised to rinse with 1 and half teaspoon of this cocktail 3 times a day for 2 minutes for the period of 8 weeks and do not eat or drink anything 30 minutes after its use. Study group will also advised to apply triamcinolone orabase containing 0.1% triamcinolone on lesions 3 times a day for the period of 8 weeks. The control group will be advised to apply only triamcinolone orabase 3 times a day for 8 weeks with the same protocol. Assessment of dimension of lesions, color, pain and burning sensation and improvement of lesions and symptoms will be done at baseline and after 4 and 8 weeks.

   Statistical Analysis The data will be coded and entered using SPSS ver 20. All the numerical variables will be presented as mean and standard deviation while the categorical variables will be reported as frequencies and percentages. the comparison of efficacy between two groups will be done through chi-square test.

   For all analysis a p-value of > 0.05 will be considered significant with a confidence level of 95%

   Ethical Considerations:

   Patients fulfilling the inclusion criteria will be informed about the aim of study, risks, benefits and a consent form will be signed by them. Study will be approved by Institutional Review Board (IRB), The University of Faisalabad.

ELIGIBILITY:
Inclusion Criteria:

- 1. Histopathologically proven patients of OLP of all age groups complaining of symptoms such as pain, burning sensitivity to hot and spicy food.

2. Who have signed informed consent.

Exclusion Criteria:

- 1. Patients who have taken any medication for OLP within 4 weeks before the start of study.

2. Pregnant and lactating women. 3. History of lichenoid reactions to beta blockers, dapsone, oral hypoglycemics, NSAIDS, pencillamine, phenothiazines, sulfonylureas, gold salts or amalgam fillings.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
healing of lesions | 6 bmonths
  healing of oral lichen planus lesions

CONTACTS AND LOCATIONS:
Overall Officials: Saima Chaudhry, PhD, Study Director — Co-coordinator
Locations (1):
- The university of Faisalabad, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No